CLINICAL TRIAL: NCT06112899
Title: The Effects of Swedish Massage and Manual Lymph Drainage After Muscle Fatigue in Healthy Young Men
Brief Title: The Effects of Swedish Massage and Manual Lymph Drainage on Muscle Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Hümeyra Kiloatar, Asst. Prof. Dr., Kutahya Health Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/02-02
Record Dates: First submitted 2023-10-23; First posted 2023-11-02 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Muscle Soreness
Keywords: Manual lympatic Drainage; Swedish Massage; Muscle Soreness
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Young Men (Experimental)
  Interventions: Behavioral: Nordic Hamstring Exercise

INTERVENTIONS:
Behavioral: Nordic Hamstring Exercise — The NHE, also referred to as the nordic curl, is designed to improve eccentric strength of the hamstring muscles. Individuals start in a kneeling position, with the torso from the knees upward held rigid and straight. The training partner ensures that the individual's feet are in contact with the ground throughout the exercise by applying pressure to the player's heels/lower legs. The individual then lowers his upper body to the ground, as slowly as possible to maximize loading in the eccentric phase. Hands and arms are used to break his forward fall and to push him back up after the chest has touched the ground, to minimize loading in the concentric phase.The exercise protocol is planned as 5 sets of 8 repetitions and 2 minutes of rest between each set.

SUMMARY:
12 healthy men aged 18-30 will be included in the study. Participants will be selected from students who regularly train and do active sports at the Faculty of Sports Sciences. All participants will do nordic hamstring exercise. Participants will rest for 20 minutes after the Nordic hamstring exercise protocol in the first week. In the second week, manual lymph drainage covering the lower extremities will be applied for 20 minutes after exercise. In the third week, a Swedish massage covering the lower extremities will be applied after exercise. The exercise protocol is planned as 5 sets of 8 repetitions and 2 minutes of rest between each set. The evaluations of the participants will be repeated 3 times: just before the test, after the test and after the application.

ELIGIBILITY:
Inclusion Criteria:

* Being male between the ages of 18-30
* Doing sports and training regularly
* Not exercising until 1 week before the study

Exclusion Criteria:

* Having a previous lower extremity injury
* Having a neurological problem that prevents exercise
* Does not have a diagnosed cardiovascular problem

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Lactic Acid Level | through study completion, an average of 1 year
  Blood lactate levels will be measured using a portable lactic acid analyzer (Lactate Scout+, SensLab GmbH, Leipzig, Germany), which can measure electroenzymatically in approximately 15 seconds from a drop of capillary blood sample taken from the fingertip. Blood samples will be taken using a lancet gun (Vital Plus, China). Before the evaluation, the patient's fingertip will be wiped with alcohol cotton and allowed to dry. Before all measurements, the analyzer will be calibrated with control solutions of known concentration according to the manufacturer's instructions.
Gait and Balance | through study completion, an average of 1 year
  Participants' walking parameters will be measured and recorded instantly with the Zebris™ FDM-2 device. The data obtained from the device will be recorded and compiled into a report via Zebris software installed on the computer. Participants will be asked to walk at least 8 steps on the walking platform at a pace they feel comfortable with. Step length, step width, number of steps per minute (cadence), walking speed (m/s), symmetry of center of pressure changes during walking (length of walking line, length of contact line of each step), maximum power on the feet during walking (N/cm2). ). Participants will be asked to stand with their arms hanging at their sides and their eyes fixed on a point 3 meters away in front of them, maintaining their posture as much as possible for 60 seconds. The changes in the center of pressure (ellipse area (mm2)), the total load on the right and left feet, and the anteroposterior foot distribution will be obtained.
Jumping Performance | through study completion, an average of 1 year
  Jumping performance will be evaluated with the OptoJump (Microgate, Italy) device. Using the system software, a profile will be created for each participant and BFS Vertical Jump, acoustic reaction and stiffness will be selected from the test protocols in the system.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendiguchia J, Arcos AL, Garrues MA, Myer GD, Yanci J, Idoate F. The use of MRI to evaluate posterior thigh muscle activity and damage during nordic hamstring exercise. J Strength Cond Res. 2013 Dec;27(12):3426-35. doi: 10.1519/JSC.0b013e31828fd3e7. PMID 23524362
- [Background] Poppendieck W, Wegmann M, Ferrauti A, Kellmann M, Pfeiffer M, Meyer T. Massage and Performance Recovery: A Meta-Analytical Review. Sports Med. 2016 Feb;46(2):183-204. doi: 10.1007/s40279-015-0420-x. PMID 26744335
- [Background] Cairns SP. Lactic acid and exercise performance : culprit or friend? Sports Med. 2006;36(4):279-91. doi: 10.2165/00007256-200636040-00001. PMID 16573355